CLINICAL TRIAL: NCT00476632
Title: Epidemiology Controls Using Healthy Participants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0112; P50CA100632 (NIH); 5R01CA070917-08 (NIH)
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Epidemiology; Questionnaire; Controls
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 ½ tablespoons of blood drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control: Person with no history of cancer.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 50 Minute Interview
  Other Names: Survey

SUMMARY:
The goal of this research study is to identify biologic and lifestyle factors that may increase a person's risk of developing certain types of cancer.

DETAILED DESCRIPTION:
For this study, you will be asked to complete a personal interview. During the interview, you will be asked questions about your demographics (age, sex, etc.), certain environmental exposures, your medical history, family history, your diet, and your smoking and alcohol use histories. It should take around 50 minutes to complete the interview.

You will also have around 2 ½ tablespoons of blood drawn for special tests. These tests will look for any biologic factors associated with certain cancers. The interview and blood draw will be scheduled at the time and place of your convenience. You will not be informed of the results of any of the testing done with your samples.

There is a possibility that you might be contacted in the future about if researchers need clarification on any of information already collected. You are free to refuse any further participation if you wish.

This is an investigational study. Up to 1,500 participants will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ages 18 and over with no prior cancer
2. Willing and able to complete an administered questionnaire
3. Willing and able to donate 30 mL of blood

Exclusion Criteria:

1. Individuals with prior cancer
2. Individuals under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years or older with no history of cancer.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2004-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To identify biologic and lifestyle factors that may increase a person's risk of developing certain types of cancer. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Daniel-MacDougall, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org